CLINICAL TRIAL: NCT04072237
Title: Phase 1 Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Ascending Doses of Subcutaneous Marzeptacog Alfa (Activated) in Adult Subjects With Hemophilia
Brief Title: Study of Coagulation Faction VIIa Variant Marzeptacog Alfa (Activated) in Adult Subjects With Hemophilia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MAA-102
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Hemophilia A; Hemophilia B; Hemophilia A With Inhibitor; Hemophilia B With Inhibitor; Hemophilia A Without Inhibitor; Hemophilia B Without Inhibitor
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — marzeptacog alfa (activated)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): MarzAA (Coagulation Factor VIIa variant) 18 µg/kg intravenously (Stage 1) followed by MarzAA 30 µg/kg subcutaneously (SC) (Stage 2), MarzAA 45 µg/kg SC (Stage 3), MarzAA 60 µg/kg SC (Stage 4), MarzAA 2x30 µg/kg SC (Stage 5), MarzAA 90 µg/kg SC (Stage 6), MarzAA 120 µg/kg SC (Stage 7), MarzAA 2×60 µg/kg SC (Stage 8), MarzAA 3x60 µg/kg SC (Stage 9)
  Interventions: Biological: MarzAA (marzeptacog alfa [activated])

INTERVENTIONS:
Biological: MarzAA (marzeptacog alfa [activated]) — Single intravenous dose and ascending doses of subcutaneous injection of MarzAA (Coagulation Faction VIIa Variant)

SUMMARY:
This multi-center, open label Phase 1 study will evaluate the pharmacokinetics, pharmacodynamics, and safety of a single IV dose of MarzAA followed by ascending single SC doses of MarzAA in adult subjects with moderate or severe Hemophilia A or B, with or without an inhibitor.

DETAILED DESCRIPTION:
This multi-center, open label Phase 1 study will evaluate the pharmacokinetics, pharmacodynamics, and safety of a single IV dose of MarzAA followed by ascending single SC doses of MarzAA in adult subjects with moderate or severe Hemophilia A or B, with or without an inhibitor. The study will enroll at least 8 adult male subjects with moderate or severe Hemophilia A or B with or without an inhibitor, in each dosing stage. Each subject will receive escalating doses of MarzAA for each stage of the study (except for Stage 5, where subjects receive the same dose as in Stage 4 split between two anatomical sites).

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe congenital Hemophilia A or B, with or without an inhibitor
* Male, age 18 or older
* Affirmation of informed consent with signature confirmation before any trial related activities

Exclusion Criteria:

* Inability to discontinue and washout prophylaxis treatment 72 hours prior to dosing.
* Previous participation in a trial involving SC Administration of rFVIIa or any trial using a modified amino-acid sequence FVIIa
* Known positive antibody to FVII or FVIIa detected by central laboratory at screening
* Have a coagulation disorder other than hemophilia A or B, with or without an inhibitor
* Significant contraindication to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, PhD, MMM, Study Director — Sponsor GmbH
Locations (5):
- Bulgaria (2):
  - Medical Center "Hippocrates - N", Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
- Russia (3):
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - National Medical Hematology Research Center, Moscow
  - Municipal Policlinic # 37, City Center for Hemophilia Treatment, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No
This is an open label study so each investigator will have full access to all study subject data that is entered into the database.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fourteen subjects were screened in the study and three subjects were screen failures. Two subjects failed due to having a known positive antibody at screening, and one subject failed screening due to other.
Groups:
- Overall Study Population: Coagulation Factor VIIa variant: Single intravenous dose and ascending doses of subcutaneous injection of MarzAA
Period: Stage I: MarzAA 18 µg/kg IV
Arm/Group | Overall Study Population
Started | 11
Completed | 10
Not Completed | 1
Period: Stage 2: MarzAA 30 µg/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 3: MarzAA 45 µg/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 4: MarzAA 60 µg/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 5: MarzAA 2 x 30 ug/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 6: MarzAA 90 µg/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 7: MarzAA 120 µg/kg SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 8: MarzAA 2 x 60 µg/kg Q3H SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0
Period: Stage 9: MarzAA 3 x 60 µg/kg Q3H SC
Arm/Group | Overall Study Population
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: MarzAA (Marzeptacog Alfa [activated], Coagulation Factor VIIa variant) 18 µg/kg intravenously (Stage 1) followed by MarzAA 30 µg/kg subcutaneously (SC) (Stage 2), MarzAA 45 µg/kg SC (Stage 3), MarzAA 60 µg/kg SC (Stage 4), MarzAA 2x30 µg/kg SC (Stage 5), MarzAA 90 µg/kg SC (Stage 6), MarzAA 120 µg/kg SC (Stage 7), MarzAA 2×60 µg/kg SC (Stage 8), MarzAA 3x60 µg/kg SC (Stage 9)
Arm/Group | Study Population
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Bulgaria | 8
  Russia | 3

OUTCOME MEASURES:

1. Primary Outcome: Comparative MarzAA Activity by Dose Level/Stage - AUC0-∞ and AUC0-last
Description: Comparative pharmacokinetics (PK) by dose level/stage based on examination of AUC frequencies of these for each of the dose groups
Time Frame: Dosing period for each stage was approximately 3 days, with a maximum of approximately 8 weeks of dosing, depending on participation in all 9 stages and time elapsed between each study stage.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Stage 1 MarzAA 18 µg/kg IV: Single intravenous dose of MarzAA, coagulation factor VIIa variant
- Stage 2 MarzAA 30 µg/kg SC; Stage 3 MarzAA 45 µg/kg SC; Stage 4 MarzAA 60 µg/kg SC; Stage 6 MarzAA 90 µg/kg SC; Stage 7 MarzAA 120 µg/kg SC: Single subcutaneous injection of MarzAA, coagulation factor VIIa variant
- Stage 5 MarzAA 2×30 µg/kg SC: Two subcutaneous injections of MarzAA, coagulation factor VIIa variant
- Stage 8 2×60 µg/kg SC Q3H: Two subcutaneous injections of MarzAA, coagulation factor VIIa variant, every 3 hours
- Stage 9 3×60 µg/kg SC Q3H: Three subcutaneous injections of MarzAA, coagulation factor VIIa variant, every 3 hours
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
h*ng/mL
  AUC0-∞ | 1390.0 (433.99) | 516.4 (170.01) | 849.4 (275.00) | 1060.0 (205.86) | 1025.6 (328.31) | 1487.9 (429.39) | 2087.6 (648.85) | 2108.0 (409.00) | 3235.5 (735.43)
  AUC0-last | 1382.6 (431.45) | 429.5 (178.30) | 692.9 (232.53) | 922.1 (192.38) | 934.1 (305.32) | 1322.6 (440.03) | 1868.1 (651.04) | 1939.1 (357.25) | 3038.1 (760.56)

2. Primary Outcome: Comparative MarzAA Activity by Dose Level/Stage - AUCT1-T2 Normalized by Dose = AUC0-last/Dose
Description: Comparative pharmacokinetics by dose level/stage based on examination of AUC frequency of these for each of the dose groups
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*kg/mL
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
h*kg/mL | 76.81 (23.97) | 14.32 (5.94) | 15.40 (5.17) | 15.37 (3.206) | 15.57 (5.09) | 14.70 (4.89) | 15.57 (5.43) | 16.16 (2.98) | 16.88 (4.23)

3. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - Cmax
Description: Change in Cmax at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL | 419.49 (185.18) | 18.96 (10.29) | 32.91 (18.49) | 41.88 (15.24) | 40.75 (15.98) | 54.29 (24.68) | 76.70 (34.51) | 68.04 (26.58) | 98.33 (32.64)

4. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - Tmax
Description: Change in Tmax at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hour | 0.17 (0.29) | 7.50 (1.60) | 7.38 (2.56) | 8.25 (1.39) | 6.75 (1.398) | 7.12 (1.55) | 8.25 (1.39) | 8.37 (2.67) | 12.25 (5.04)

5. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - T1/2eqα
Description: Change in T1/2eqα at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours | 1.73 (0.55) | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose. | NA (NA) — T1/2eqα was measured and derived only at IV dose.

6. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - T1/2λ-z
Description: Change in T1/2λ-z at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours | 3.3 (0.38) | 18.55 (5.88) | 19.26 (6.69) | 15.70 (3.45) | 13.05 (5.07) | 15.50 (5.65) | 15.03 (4.43) | 18.82 (5.82) | 18.07 (6.78)

7. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - CL
Description: Change in CL at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mL/h | 14.22 (4.66) | 63.33 (19.64) | 57.85 (18.21) | 58.88 (13.68) | 63.92 (20.36) | 65.13 (18.67) | 64.39 (26.93) | 59.05 (12.68) | 58.22 (13.28)

8. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - Vd1
Description: Change in Vd1 at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mL | 53.41 (18.02) | 1868.28 (962.02) | 1651.05 (799.32) | 1400.41 (478.92) | 1344.19 (557.26) | 1577.63 (791.28) | 1509.24 (796.50) | 1699.49 (474.39) | 1717.33 (629.45)

9. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - BAabs
Description: Change in BAabs at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Percentage | 100 (100) | 19.47 (8.07) | 21.52 (10.63) | 21.32 (7.42) | 20.87 (6.32) | 19.84 (7.20) | 21.24 (9.32) | 23.00 (8.98) | 23.32 (6.69)

10. Secondary Outcome: Comparative MarzAA Activity of Intravenous and Subcutaneous - Mean Residence Time
Description: Change in Mean Residence Time at each stage for each dose group
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours | 3.77 (0.42) | 28.25 (9.18) | 28.10 (9.94) | 23.79 (5.40) | 20.96 (5.58) | 23.42 (7.47) | 22.80 (5.9211) | 29.04 (7.88) | 29.32 (8.60)

11. Secondary Outcome: Effect of Split Injections on MarzAA Activity by Dose Level/Stage - AUC From T1 to T2 Norm by Dose
Description: PK analysis by route of administration, dose level/stage of the study based on examination of AUC for each of the dose groups.
  Split dose (2*30 µg/kg) vs. (60 µg/kg)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*kg/mL
Groups:
- Stage 4 MarzAA 60μg/kg SC: Single subcutaneous injection of MarzAA, coagulation factor VIIa variant
- Stage 5 MarzAA 2×30μg/kg SC: Two subcutaneous injections of MarzAA, coagulation factor VIIa variant
Arm/Group | Stage 4 MarzAA 60μg/kg SC | Stage 5 MarzAA 2×30μg/kg SC
Number analyzed (Participants) | 8 | 8
h*kg/mL | 15.3687 (3.20630) | 15.5688 (5.08859)

12. Secondary Outcome: Effect of Split Injections on MarzAA Activity by Dose Level/Stage - AUC Infinity Obs and AUC to Last Nonzero Conc
Description: as for outcome 11
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Stage 4 MarzAA 60μg/kg SC: Single subcutaneous injection of MarzAA coagulation factor VIIa variant
- Stage 5 MarzAA 2×30μg/kg SC: Two subcutaneous injections of MarzAA coagulation factor VIIa variant
Arm/Group | Stage 4 MarzAA 60μg/kg SC | Stage 5 MarzAA 2×30μg/kg SC
Number analyzed (Participants) | 8 | 8
h*ng/mL
  AUC Infinity Obs | 1060.0 (205.86) | 1025.6 (328.31)
  AUC to Last Nonzero Conc | 922.1 (192.38) | 934.1 (305.32)

13. Secondary Outcome: Change in Coagulation Parameters - Prothrombin Time (PT)
Description: Maximum change in PT from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-7 (SC).
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Stage 1 MarzAA 18 µg/kg SC: Single intravenous dose of MarzAA, coagulation factor VIIa variant
Arm/Group | Stage 1 MarzAA 18 µg/kg SC | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
seconds | -1.36 (0.57) | -1.41 (0.86) | -1.16 (0.68) | -1.09 (0.58) | -1.29 (0.86) | -1.07 (0.79) | -1.37 (0.54) | -1.36 (0.60) | -1.35 (0.62)

14. Secondary Outcome: Change in Coagulation Parameters - Activated Partial Thromboplastin Time (aPTT)
Description: Maximum change in aPTT from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stage 1 MarzAA 18 µg/kg SC | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
seconds | -11.69 (3.71) | 1.91 (3.21) | -2.33 (4.28) | -2.18 (2.63) | -2.51 (2.09) | -2.85 (1.82) | -2.10 (3.02) | -2.92 (3.01) | -5.13 (2.59)

15. Secondary Outcome: Change in Coagulation Parameters - Thrombin Generation Time (TGT) - TGT-Peak
Description: Maximum change in TGT parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
nM | 64.0 (65.32) | 14.9 (31.69) | 28.3 (21.04) | 42.3 (32.13) | 45.4 (30.84) | 33.0 (25.16) | 44.3 (46.10) | 45.6 (19.18) | 41.3 (30.47)

16. Secondary Outcome: Change in Coagulation Parameters - Thrombin Generation Time (TGT) - TGT-Lag and TGT-Time to Peak
Description: Maximum change in TGT parameters from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Stage 5 MarzAA 2×30 µg/kg SC: Two single subcutaneous injections of MarzAA, coagulation factor VIIa variant
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
minutes
  TGT-Lag | -1.30 (1.231) | -1.21 (0.613) | -1.11 (0.391) | -1.42 (0.645) | -1.38 (0.311) | -1.07 (0.655) | -1.33 (0.396) | -1.54 (0.507) | -1.13 (0.688)
  TGT-Time to Peak | -3.88 (3.302) | -2.22 (2.309) | -2.76 (1.226) | -3.53 (2.313) | -3.68 (1.290) | -3.73 (1.926) | -3.73 (2.024) | -3.70 (1.681) | -3.25 (1.756)

17. Secondary Outcome: Change in Coagulation Parameters - Thrombin Generation Time (TGT) - TGT-Endogenous Thrombin Potential
Description: Maximum change in TGT parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: nM•minutes
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
nM•minutes | 215.9 (337.55) | 158.6 (247.55) | 94.3 (148.51) | 149.5 (256.34) | 211.0 (190.22) | 133.0 (193.85) | 216.9 (184.54) | 164.6 (58.49) | -187.3 (474.61)

18. Secondary Outcome: Change in Thrombogenicity Parameter - Fibrinogen
Description: Maximum change in thrombogenicity parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mg/dL | -13.2 (23.83) | 13.3 (29.65) | -23.6 (34.04) | 16.0 (37.67) | 7.6 (51.69) | -31.0 (42.02) | 21.6 (56.61) | -12.5 (32.74) | -8.0 (33.72)

19. Secondary Outcome: Change in Thrombogenicity Parameter - Prothrombin Fragments 1 + 2
Description: Maximum change in thrombogenicity parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
pmol/L | 1903.5 (3809.47) | 206.3 (545.97) | 56.0 (158.02) | 76.5 (118.78) | 383.9 (324.41) | 974.5 (2407.09) | 1744.9 (4367.48) | 236.5 (459.58) | 284.9 (672.80)

20. Secondary Outcome: Change in Thrombogenicity Parameter - Thrombin/Antithrombin
Description: Maximum change in thrombogenicity parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
µg/L | 105.09 (254.951) | 62.34 (156.899) | 10.41 (19.586) | 63.57 (181.409) | 138.19 (202.946) | 56.79 (146.603) | 10.46 (15.648) | 18.90 (38.191) | 3.75 (3.231)

21. Secondary Outcome: Change in Thrombogenicity Parameter - D-Dimer
Description: Maximum change in thrombogenicity parameter from pre-dose
Time Frame: From predose to Day 2 at stage 1 (IV). From predose to Day 3 at stages 2-9 (SC).
Measure: Mean (Standard Deviation); unit: mg/L Fibrinogen Equivalent Unit
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
mg/L Fibrinogen Equivalent Unit | 0.141 (0.214) | -0.054 (0.104) | 0.110 (0.080) | 0.039 (0.073) | 0.285 (0.605) | 0.200 (0.175) | 0.211 (0.285) | 0.111 (0.125) | 0.256 (0.173)

22. Secondary Outcome: Occurrence of an Antibody Response to MarzAA
Description: Occurrence of an antibody response to MarzAA and whether it is inhibitory and cross-reactive to wild-type recombinant coagulation FVII (wt-rFVII) or wt-FVIIa
Time Frame: From time of first dose of MarzAA until date of first occurrence of clinical event, assessed up to End of Study. Dosing period for each stage was approximately 3 days, with a maximum of approximately 8 weeks of dosing.
Measure: Number; unit: participants with an occurrence
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg SC Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
participants with an occurrence | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Occurrence of Clinical Thrombotic Event
Description: Occurrence of clinical thrombotic event not attributable to another cause
Time Frame: From the date of first dose of MarzAA until date of first occurrence of clinical event, assessed up to End of Study. Dosing period for each stage was approximately 3 days, with a maximum of approximately 8 weeks of dosing.
Measure: Number; unit: participants with an occurrence
Groups:
- Stage 9 3×60 µg/kg Q3H: Three subcutaneous injections of MarzAA, coagulation factor VIIa variant, every 3 hours
Arm/Group | Stage 1 MarzAA 18 µg/kg IV | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 2×60 µg/kg SC Q3H | Stage 9 3×60 µg/kg Q3H
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
participants with an occurrence | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were defined as any event that either began or worsened after the first administration of study drug and within 28 days of the last dose.
Description: An adverse event (AE) was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related.
  An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug, without any judgment about causality. An AE could arise from any use of the drug (eg, off label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.
Groups:
- Stage 1 MarzAA 18 µg/kg SC: Single intravenous dose of MarzAA
- Stage 2 MarzAA 30 µg/kg SC; Stage 3 MarzAA 45 µg/kg SC; Stage 4 MarzAA 60 µg/kg SC; Stage 6 MarzAA 90 µg/kg SC; Stage 7 MarzAA 120 µg/kg SC: Single subcutaneous injection of MarzAA
- Stage 5 MarzAA 2×30 µg/kg SC: Two subcutaneous injections of MarzAA
- Stage 8 MarzAA 2×60 µg/kg SC Q3H: Two subcutaneous injections of MarzAA every 3 hours
- Stage 9 MarzAA 3×60 µg/kg SC Q3H: Three subcutaneous injections of MarzAA every 3 hours
Arm/Group | Stage 1 MarzAA 18 µg/kg SC | Stage 2 MarzAA 30 µg/kg SC | Stage 3 MarzAA 45 µg/kg SC | Stage 4 MarzAA 60 µg/kg SC | Stage 5 MarzAA 2×30 µg/kg SC | Stage 6 MarzAA 90 µg/kg SC | Stage 7 MarzAA 120 µg/kg SC | Stage 8 MarzAA 2×60 µg/kg SC Q3H | Stage 9 MarzAA 3×60 µg/kg SC Q3H
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 3/8 | 0/8 | 1/8 | 1/8 | 0/8 | 2/8 | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 MarzAA 18 µg/kg SC (N=11) | Stage 2 MarzAA 30 µg/kg SC (N=8) | Stage 3 MarzAA 45 µg/kg SC (N=8) | Stage 4 MarzAA 60 µg/kg SC (N=8) | Stage 5 MarzAA 2×30 µg/kg SC (N=8) | Stage 6 MarzAA 90 µg/kg SC (N=8) | Stage 7 MarzAA 120 µg/kg SC (N=8) | Stage 8 MarzAA 2×60 µg/kg SC Q3H (N=8) | Stage 9 MarzAA 3×60 µg/kg SC Q3H (N=8)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04072237/Prot_SAP_000.pdf